CLINICAL TRIAL: NCT02169778
Title: Effect of Intermittent Versus Continuous Energy Restriction on Compensatory Mechanisms Activated During Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Monash University (Other); Portuguese Research Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/754
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Weight loss; Intermittent energy restriction; Metabolic compensation; Diet therapy
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent energy restricted diet (Experimental): The intermittent energy restricted group will undergo 3 nonconsecutive days of partial fasting per week. During the 3 days of partial fasting, participants will be asked to consume a very-low calorie diet (VLCD) providing 550kcal/day for women and 650kcal/day for men. The VLCD products provide 110kcal/pack and include a variety of shakes, smoothies and soups. For the feeding days a diet matching energy needs will be prescribed, using meal replacements (such as smoothies, soups and cereal bars) and conventional food. Drinking at least 2.5 liters of non-caloric liquids will be recommended.
  Interventions: Behavioral: Intermittent energy restricted diet
- Continuous energy restricted diet (Experimental): The continuous energy restricted group will be prescribed a low calorie diet (LCD) with 33% energy restriction, using meal replacements (such as smoothies, soups and cereal bars) and conventional food. The diets' macronutrient composition of the two groups will be matched (50% carbohydrates, 20% protein and 30% fat).
  Interventions: Behavioral: Continuous energy restricted diet

INTERVENTIONS:
Behavioral: Intermittent energy restricted diet
  Arms: Intermittent energy restricted diet
Behavioral: Continuous energy restricted diet
  Arms: Continuous energy restricted diet

SUMMARY:
Obesity has become a global epidemic with huge public health implications. Although clinical significant weight loss can be achieved by a combination of diet and behavioral modification, strong metabolic adaptations, with increased appetite and suppressed energy expenditure, are activated, which compromise weight loss maintenance and increase the risk of relapse. The aim of this project is to compare the effects of intermittent versus continuous energy restriction on the compensatory responses previously described using two low calory diets, with a similar macronutrient distribution. More specifically, this study will analyze, in the short-term, if an intermittent energy restricted diet is associated with less appetite and low reduction in energy expenditure when compared with a continuous energy restricted diet. This project can bring large practical benefits concerning the design of weight loss programs to minimize weight relapse.

ELIGIBILITY:
Inclusion Criteria:

* adult (18-50 years old)
* obese healthy volunteers (30<BMI<40 kg/m2)
* weight stable on the last three months (<2kg), not currently dieting to lose weight and with an inactive lifestyle

Exclusion Criteria:

* history of endocrine/cardiovascular/pulmonary/kidney disease
* anaemia
* milk intolerance
* depression or other psychological disorders
* eating disorders
* drug or alcohol abuse within the last two years
* current medication known to affect appetite or induce weight loss
* a planned surgery during the study period
* participating in another research study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Appetite related hormones | 12 weeks after the intervention
  Appetite-related hormones (active Ghrelin, PYY, GLP-1, CCK) will be measured in fasting and every 30 minutes up to 2,5 hours.

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | 12 weeks after the intervention
  RMR measured by indirect calorimetry
Exercise efficiency | 12 weeks after the intervention
  Exercise efficiency measured by graded exercise on a bike
Body composition | 12 weeks after the intervention
  RMR measured by indirect calorimetry
Body composition | At 6 months from baseline
  RMR measured by indirect calorimetry
Body composition | At 1 year from baseline
  RMR measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Coutinho SR, Halset EH, Gasbakk S, Rehfeld JF, Kulseng B, Truby H, Martins C. Compensatory mechanisms activated with intermittent energy restriction: A randomized control trial. Clin Nutr. 2018 Jun;37(3):815-823. doi: 10.1016/j.clnu.2017.04.002. Epub 2017 Apr 7. PMID 28446382
- [Derived] Castela I, Rodrigues C, Ismael S, Barreiros-Mota I, Morais J, Araujo JR, Marques C, Silvestre MP, Angelo-Dias M, Martins C, Borrego LM, Monteiro R, Coutinho SR, Calhau C, Faria A, Pestana D, Martins C, Teixeira D. Intermittent energy restriction ameliorates adipose tissue-associated inflammation in adults with obesity: A randomised controlled trial. Clin Nutr. 2022 Aug;41(8):1660-1666. doi: 10.1016/j.clnu.2022.06.021. Epub 2022 Jun 18. PMID 35772219
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717